CLINICAL TRIAL: NCT00950820
Title: An Open-label Randomized Phase II Study of Panitumumab Plus Oral Capecitabine and Infusional Oxaliplatin (XELOX) or XELOX Alone for Second-line Treatment of Patients With Metastatic Colorectal Cancer (VOXEL-Study)
Brief Title: Study to Evaluate the Effects of Panitumumab if Combined With Chemotherapy for 2nd Treatment of Colorectal Cancer
Acronym: VOXEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment rate to low; changed environment made protocol in its current state obsolete
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO KRK 0107
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Neoplasms
Keywords: Open-label; Phase-II-Study; Randomized; Metastatic; Colorectal; Cancer; Panitumumab; Vectibix®; second-line-treatment; KRAS
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Oxaliplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Panitumumab + XELOX (Experimental): KRAS mutational status wild-type: Panitumumab plus Oxaliplatin and Capecitabine (XELOX)
  Interventions: Drug: Oxaliplatin, Capecitabine, Panitumumab
- XELOX (KRAS mutational status wt) (Other): KRAS mutational status wild-type: Oxaliplatin and Capecitabine (XELOX)
  Interventions: Drug: Oxaliplatin, Capecitabine
- XELOX (KRAS mutational status mutant) (Other): KRAS mutational status mutant: Oxaliplatin and Capecitabine (XELOX)
  Interventions: Drug: Oxaliplatin, Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin, Capecitabine, Panitumumab — Panitumumab at a dose of 9 mg/kg BW every three weeks will be administered on day 1 of each cycle just prior to administration of chemotherapy.
  The XELOX regimen is defined as a 2 hour infusion of oxaliplatin 130 mg/m² on day 1 followed by capecitabine 1000 mg/m² bid per os. Capecitabine administration will commence on the evening of day 1 and complete after the morning dose on day 15.
  Arms: Panitumumab + XELOX
Drug: Oxaliplatin, Capecitabine — The XELOX regimen is defined as a 2 hour infusion of oxaliplatin 130 mg/m² on day 1 followed by capecitabine 1000 mg/m² bid per os. Capecitabine administration will commence on the evening of day 1 and complete after the morning dose on day 15.
  Arms: XELOX (KRAS mutational status mutant); XELOX (KRAS mutational status wt)

SUMMARY:
The purpose of this interventional study is to investigate whether there is evidence that panitumumab in combination with XELOX (capecitabine plus oxaliplatin) chemotherapy will safely increase progression-free survival, above that of XELOX alone in subjects with KRAS wild-type metastatic colorectal cancer who have not responded to or progressed after first line therapy with irinotecan and a fluoropyrimidine.

Further Objectives Exploratory objectives may include investigation of potential correlations between the treatment regimen and epidermal growth factor receptor (EGFR) expression, detection of the functional genetic polymorphisms of the EGFR gene, EGFR gene amplification (FISH), EGFR downstream protein and gene expression parameters, proteomics and epigenetics.

DETAILED DESCRIPTION:
Subjects with metastatic colorectal cancer with KRAS-wildtype will be randomized in a 1:1 ratio to receive a 2nd line treatment regimen of panitumumab plus oxaliplatin and capecitabine (XELOX) or XELOX alone. Before randomization tumour of all subjects will be analyzed to detect the KRAS mutational status. Subjects will only be randomized into these two arms if the tumour shows KRAS wild-type. Subjects with KRAS mutant colorectal tumours will receive XELOX alone. Subjects will receive treatment cycles every three weeks. Treatment will continue until subjects are diagnosed with disease progression or intolerable toxicity, at which time the subjects will be withdrawn from the treatment phase. If a subject withdraws from chemotherapy due to toxicity the subjects will be allowed to continue with panitumumab monotherapy with or without one of the chemotherapy components until disease progression. After withdrawing panitumumab and XELOX treatment, all subjects will end the treatment phase and will enter a follow-up phase until 6 months after the last patient stopped treatment (with a safety follow-up visit after 56 days ± 3 days and long term follow-up visits every 12 weeks). During the treatment phase subjects will be evaluated for tumour response every 9 weeks (± one week) through to week 45, and every 12 weeks (± two weeks) thereafter, until disease progression. Subjects with symptoms suggestive of disease progression should be evaluated for tumour response at the time symptoms occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or more, with histologically or cytologically-confirmed and radiologically-measurable metastatic colorectal cancer.
* One prior chemotherapy regimen for mCRC consisting of first-line fluoropyrimidine and irinotecan based chemotherapy. Subjects must have disease progression (as assessed by the investigator) and must be no candidates for primary metastasectomy.
* Measurable disease according to RECIST 1.1 guidelines. All sites of disease must have been evaluated within 28 days prior to registration / randomization, and diagnosed by the investigator.
* Liver and kidney function within defined ranges and sufficient bone marrow reserve.

Exclusion Criteria:

* Central nervous system metastases, or significant cardiovascular disease.
* Prior anti-EGFR antibody therapy (e.g. cetuximab) or treatment with small molecule EGFR tyrosine kinase inhibitors (e.g. erlotinib).
* Prior treatment with oxaliplatin for metastatic disease. Adjuvant therapy with oxaliplatin based combination for non-metastatic disease is allowed if terminated > 6 months prior to initiation of screening and without progression during the treatment with oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months for subjects with KRAS wild-type tumours | 6 months

SECONDARY OUTCOMES:
PFS | end of study
Objective-response-rate | end of study
Disease-control-rate | end of study
Time-to-response | end of study
time-to-progression | end of study
duration-of-stable-disease | end of study
time-to-treatment-failure | end of study
overall-survival | end of study
safety-endpoints | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Grunewald, PD Dr., Principal Investigator — Gemeinschaftspraxis Hämatologie / Onkologie Im Prüfling 17-19 60389 Frankfurt
Locations (1):
- AIO-Studien-gGmbH, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Related Info — http://www.aio-portal.de